CLINICAL TRIAL: NCT01748617
Title: The Potential for Pomegranate Juice to Ameliorate Endothelial Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janet Novotny (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Janet Novotny, Principal Investigator, USDA Beltsville Human Nutrition Research Center
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: HS41
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pomegranate Juice (Experimental): Acute ingestion of pomegranate juice with high fat meal.
  Interventions: Other: Controlled diet
- Control (Placebo Comparator): Acute ingestion of juice-free sweetened beverage with high fat meal.
  Interventions: Other: Controlled diet

INTERVENTIONS:
Other: Controlled diet — 1 week of controlled diet

SUMMARY:
This study will be a randomized, double-blind, crossover intervention to investigate the health effects of acute ingestion of pomegranate juice when consumed with a high fat meal. After one week of controlled dietary intervention, subjects will consume a high fat morning meal supplemented with either pomegranate juice or a juice-free sweetened beverage. After consumption of the breakfast meal, subjects will be assessed for endothelial function and postprandial meal response.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 25-70 years
* Body mass index (BMI) ≥ 19 and ≤ 38
* Willingness and ability to make scheduled appointments at clinical site as required by study protocol

Exclusion Criteria:

* Known (self-reported) allergy or adverse reaction to study foods
* Presence of kidney disease, liver disease, gout, untreated or unstable hyperthyroidism, untreated or unstable hypothyroidism, certain cancers, gastrointestinal disease, pancreatic disease, other metabolic diseases, or malabsorption syndromes
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* Fasting triglycerides > 300 mg/dL
* Fasting glucose > 126 mg/dL
* Use of cholesterol lowering medication
* Blood pressure > 180/100 or hypertension treated with calcium channel blockers, direct acting vasodilators, or beta blockers
* Fingernails longer than 0.25 inch beyond the finger tip, or unwillingness to cut fingernails to this length during endothelial function testing
* History of bariatric or certain other surgeries related to weight control
* History of major surgery within 3 months of enrollment
* Smokers or other tobacco users (during 6 months prior to the start of the study)
* Antibiotic use during the intervention or for 3 months prior to the intervention period
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Volunteers who have lost 10% of body weight within the last 6 months
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in endothelial function | 0 hour and 3 hour
  After a consuming controlled diet for 1 week, subjects will report in the morning after a 12 hour fast. Upon arrival , subjects' endothelial function will be assessed by measuring endothelium-dependent flow mediated dilation of the peripheral bed (EndoPAT, Itamar Medical, Israel). For this test, subjects will rest in the supine position with a brachial blood pressure cuff on one arm and a finger tip probe on each of two fingers (one on the left hand, one on the right hand). After 5 minutes of rest, the blood pressure cuff will be inflated and remain inflated for 5 minutes. Then the cuff pressure will be released and the subject will remain resting for 5 additional minutes. This test will be repeated 3 hours after the test meal.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Novotny, Ph.D., Principal Investigator — USDA Beltsville Human Nutrition Research Center
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States